CLINICAL TRIAL: NCT05057338
Title: Innovative Follow-up Across Health Care Levels to Optimize Functions, Physical Activity and Employment for Individuals With MS: A Pilot Feasibility Study
Brief Title: Functions, Physical Activity and Employment for Individuals With MS: A Pilot Feasibility Study
Acronym: CoreDISTp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: Nord University (Other); Hasselt University (Other); Helse Nord (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CoreDISTparticipation
Record Dates: First submitted 2021-08-27; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Physiotherapy; neurology; MS nurse; coordination of care; balance; walking; physical activity; employment
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: RCT with two arms: intervention group and control group.
Who Masked: Outcomes Assessor
Masking Description: Assessor is masked for group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CoreDISTparticipation (Experimental): a) at the MS-OP clinic, in addition to the regular consultations, the patient will have a structured digital conversation with the MS-nurse addressing work related issues and a session with a physiotherapist exploring possibilities for change in balance and walking; b) in the municipality, a physiotherapist will continue exploration of improvements, followed by four weeks of GroupCoreDIST focusing on balance, walking and physical activity and conducted in groups of 3-5 individuals with MS and led by a physiotherapist.
  To promote participation in employment, a structured digital meeting between each patient, the MS-nurse, the patient's employer, and the physiotherapist will take place; followed by c) four weeks of outdoor group based exercises and physical activity led by a physiotherapist, complemented with an evaluation form regarding employment and physical activity.
  Interventions: Behavioral: CoreDISTparticipation
- Standard care (Active Comparator): The control group will receive the usual consultations at the MS-OP clinic including exploration of possibilities for change in balance and walking together with physiotherapist at the MS-OP clinic. The control group will furthermore follow standard care (their usual follow-up) in the municipality.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: CoreDISTparticipation — CoreDISTparticipation is a thorough intervention that contains coordination of services (physiotherapy, MS-nursing and work adaptations) between the MS-OP clinic and the municipality aiming to improve function, physical activity and employment in individuals with MS.
  Arms: CoreDISTparticipation
Behavioral: Standard care — The standard care group will follow regular consultations at the MS-outpatient clinic including a session with the physiotherapist. Furthermore, this group will follow usual care in the municipality which might include other forms of physiotherapy or physical activity. These will be registered.
  Arms: Standard care

SUMMARY:
Multiple Sclerosis (MS) is a chronic disease affecting young adults. Impaired balance, walking, reduced physical activity and participation in employment are common, however, less integrated in the health care. The researchers have developed a multidisciplinary intervention and pathway delivered across health care levels targeting the promotion of balance, walking, physical activity and participation in employment. The research team will perform a pilot feasibility Randomized Controlled Trial (RCT) and interviews to investigate the feasibility of the new intervention compared to a standard care for individuals with lower levels of disability.

DETAILED DESCRIPTION:
The study addresses core elements in the health services for individuals with MS, constituting approximately 11000 in Norway. The two-armed pilot feasibility-RCT will be performed across the MS-outpatient (MS-OP) clinic, Nordland Hospital Trust, Bodø (NLSH), and in two surrounding municipalities, including 30 employed participants who will be followed for 10-weeks. The new intervention and pathway, CoreDISTparticipation, builds on GroupCoreDIST, which is previously found effective short and long term compared to standard care. CoreDISTparticipation consists of three phases: a) at the MS-OP clinic, in addition to the regular consultations, the patient will have a structured digital conversation with the MS-nurse addressing work related issues and a session with a physiotherapist exploring possibilities for change in balance and walking; b) in the municipality, a physiotherapist will continue exploration of improvements, followed by four weeks of GroupCoreDIST for 60 minutes, 2 times per week supplemented with home exercise programs focusing on balance, walking and physical activity. The participants will have access to exercise programs on videos through an open website at Nord University to digitally support home training.

To promote participation in employment, a structured digital meeting between each patient, the MS-nurse, the patient's employer, and the physiotherapist (who leads the group trainings) will take place in phase b; followed by phase c) which include four weeks of outdoor group based exercises and physical activity led by a physiotherapist, for 60 minutes, 2 times per week supplemented with the same home exercise programs as in phase b.

Evaluation of employment and physical activity will be conducted using an evaluation form.

The control group will receive usual consultations at the MS-OP clinic, as well as a session with a physiotherapist at the MS-OP clinic, exploring possibilities for change in balance and walking. In the municipality the control group will follow standard care (their usual follow-up).

The research team will examine feasibility, preliminary between-group differences regarding balance, walking, physical activity level, health related quality of life and barriers in employment, as well as the users' experiences with participation in the CoreDISTparticipation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MS (Mc Donald's criteria), Expanded Disability Status Scale ≤3.5 (no disability-fully ambulatory with moderate disability), ≥18 years, being employed. By these criteria the study will include individuals most accessible for the intervention and who have the best prospects to maintain/improve balance, walking, physical activity and participation in employment.

Exclusion Criteria:

* Retired, pregnancy at enrolment, exacerbation within two weeks prior to enrolment and other serious conditions compromising balance, walking or work capacity.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
MS Work Difficulties Questionnaire-23 | Baseline
  How frequently individuals with MS perceive psychological/cognitive (11 items)-, physical (8 items)- and external barriers (4 items) related to their current or most recent job, and is scored by a five point scale (best score 0). (Recently translated to Norwegian).
Six-Minutes Walk Test | Baseline
  Walking distance within six minutes
MS Work Difficulties Questionnaire-23 | 5 weeks post-test
  How frequently individuals with MS perceive psychological/cognitive (11 items)-, physical (8 items)- and external barriers (4 items) related to their current or most recent job, and is scored by a five point scale (best score 0). (Recently translated to Norwegian).
Six-Minutes Walk Test | 5 weeks post-test
  Walking distance within six minutes
MS Work Difficulties Questionnaire-23 | 10 week post-test
  How frequently individuals with MS perceive psychological/cognitive (11 items)-, physical (8 items)- and external barriers (4 items) related to their current or most recent job, and is scored by a five point scale (best score 0). (Recently translated to Norwegian).
Six-Minutes Walk Test | 10 week post-test
  Walking distance within six minutes

SECONDARY OUTCOMES:
Trunk Impairment Scale Norwegian Version | Baseline
  Dynamic sitting balance, 6 items, top score 16.
Mini Balance Evaluation Systems Test | Baseline
  Pro-and reactive balance, dual task and involving sit to stand, standing and walking, 14 items on a 3 point with a top score of 28
Force Platform | Baseline
  The force platform measures control in standing: symmetry/asymmetry of weight bearing with eyes open/closed, postural sway of center of pressure, and weight transfer which all together will present an outcome for standing balance.
Activity monitors outcome 1 | Baseline
  The monitors measure Physical activity levels (inactive, light, moderate, vigorous) within 7 days
Activity monitors outcome 2 | Baseline
  The monitors measure number of steps within 7 days
European Quality of Life 5-Dimension-3 Level | Baseline
  Self-perceived health related quality of life regarding five domains, each with three items, and a Visual Analog Scale (0-100) recording perceived health.
Multiple Sclerosis Walking Scale-12 | Baseline
  Limitations in walking due to MS on 12 items with a scale 1-5, best score 12
Multiple Sclerosis Impact Scale-29 | baseline
  Self-perceived physical (13 items) and psychological (9 items) impact due to MS on health related quality of life recorded by a five point scale (best score 29)
Weight | baseline
  Self reported weight by kilogram
Height | baseline
  Self reported height by centimetre
age | baseline
  Self reported age by years
Social status | baseline
  Self reported social status; married, cohabitant, living alone
Type of multiple sclerosis | baseline
  Self reported main types: relapsing remitting, primary progressive, secondary progressive
Year of diagnosis multiple sclerosis | baseline
  Self reported by year
Medications | baseline
  Self reported by type of medications
Expanded disability status scale | baseline
  Self reported or from journal functional status at last yearly control by a neurologist
Occupation | baseline
  Self reported
Percentage of work | baseline
  Self reported percentage of work the previous month
Length of education | baseline
  Self reported choices: elementary school; high school; bachelor; masters degree; Doctor of philosophy degree
Trunk Impairment Scale Norwegian Version | 5 weeks post-test
  Dynamic sitting balance, 6 items, top score 16.
Mini Balance Evaluation Systems Test | 5 weeks post-test
  Pro-and reactive balance, dual task and involving sit to stand, standing and walking, 14 items on a 3 point with a top score of 28
Force Platform | 5 weeks post-test
  The force platform measures control in standing: symmetry/asymmetry of weight bearing with eyes open/closed, postural sway of center of pressure, and weight transfer which all together will present an outcome for standing balance.
Activity monitors outcome 1 | 5 weeks post-test
  The monitors measure Physical activity levels (inactive, light, moderate, vigorous) within 7 days
Activity monitors outcome 2 | 5 weeks post-test
  The monitors measure number of steps within 7 days
European Quality of Life 5-Dimension-3 Level | 5 weeks post-test
  Self-perceived health related quality of life regarding
Multiple Sclerosis Walking Scale-12 | 5 weeks post-test
  Limitations in walking due to MS on 12 items with a scale 1-5, best score 12
Multiple Sclerosis Impact Scale-29 | 5 weeks post-test
  Self-perceived physical (13 items) and psychological (9 items) impact due to MS on health related quality of life recorded by a five point scale (best score 29)
Percentage of work | 5 weeks post-test
  Self reported percentage of work
Trunk Impairment Scale Norwegian Version | 10 weeks post-test
  Dynamic sitting balance, 6 items, top score 16.
Mini Balance Evaluation Systems Test | 10 weeks post-test
  Pro-and reactive balance, dual task and involving sit to stand, standing and walking, 14 items on a 3 point with a top score of 28
Force Platform | 10 weeks post-test
  The force platform measures control in standing: symmetry/asymmetry of weight bearing with eyes open/closed, postural sway of center of pressure, and weight transfer which all together will present an outcome for standing balance.
Activity monitors outcome 1 | 10 weeks post-test
  The monitors measure Physical activity levels (inactive, light, moderate, vigorous) within 7 days
Activity monitors outcome 2 | 10 weeks post-test
  The monitors measure number of steps within 7 days
European Quality of Life 5-Dimension-3 Level | 10 weeks post-test
  Self-perceived health related quality of life regarding
Multiple Sclerosis Walking Scale-12 | 10 weeks post-test
  Limitations in walking due to MS on 12 items with a scale 1-5, best score 12
Multiple Sclerosis Impact Scale-29 | 10 weeks post-test
  Self-perceived physical (13 items) and psychological (9 items) impact due to MS on health related quality of life recorded by a five point scale (best score 29)
Percentage of work | 10 weeks post-test
  Self reported percentage of work

CONTACTS AND LOCATIONS:
Overall Officials: Petter Oien, PhD, Study Director — Nordlandssykehuset HF
Locations (2):
- Norway (2):
  - Bodø Municipality, Bodø
  - Physiotherapy department, Nordlandssykehuset HF, Bodø

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arntzen EC, Braaten T, Fikke HK, Normann B. Feasibility of a new intervention addressing group-based balance and high-intensity training, physical activity, and employment in individuals with multiple sclerosis: a pilot randomized controlled trial. Front Rehabil Sci. 2024 Jan 8;4:1258737. doi: 10.3389/fresc.2023.1258737. eCollection 2023. PMID 38259873